CLINICAL TRIAL: NCT00339430
Title: HLA and KIR Associations With Infectious Viral Agents in an HIV Cohort of Women (WIHS)
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999902253; 02-C-N253; NCT00897689 (obsolete NCT alias)
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2010-08-18

CONDITIONS: HIV
Keywords: Genotyping; HIV; HPV; HCV; HBV

SUMMARY:
Since the beginning of the HIV/AIDS epidemic, the number of women infected with HIV has rapidly increased and is continuing to climb. The Women's Interagency HIV Study is being conducted in several cities in the United States to learn more about how HIV affects women's lives and bodies. It will examine the role of HLA and killer immunoglobulin-like receptors (KIR) in HIV and related infections in HIV-positive and HIV-negative women. The study will determine the relationship between KIR and HLA genes and the following: the risk of HIV infection; HIV levels in the blood; incidence of AIDS; response to highly active antiretroviral therapy (HAART); and response to immunotherapy.

Approximately 3,700 women will participate. Participants will visit the clinic every 6 months for 4 years. An HIV test will be given each time to HIV-negative women. A questionnaire will also be administered. A physical examination and gynecological examination will be given. Blood, vaginal swabs, and urine will be collected for testing. A biological impedance test will determine any changes in weight, waist-to-hip ratios, and breast and total body fat. Low CD4 counts and hospitalizations for HIV are to be self-reported to study staff.

DETAILED DESCRIPTION:
The aim of the study is to examine the role of HLA and killer immunolobulin-like receptors (KIR) in the natural history of HPV, HCV, and HBV in HIV-positive and HIV-negative women. The immune response to viral infection mediated by T lymphocytes is HLA restricted, suggesting that HLA class I, and class II might be associated with risk of viral infection, persistence and disease progression. Natural killer (NK) cells are a unique group of lymphocytes involved in surveillance and killing of foreign or infected cells through a mechanism involving recognition of HLA molecules by an extremely diverse set of receptors on the NK cell surface. A major group of these receptors are the KIRs. Thus, a relationship between KIR genotype and HIV infection is biologically plausible, and requires further investigation in observational studies.

The WIHS study is a prospective study, which may allow us to answer questions relating to the role of host HLA and KIR genotype on duration of infection, and the development of virus-associated diseases such as cervical cancer (related to HPV infection), and liver cancer (HBV and HCV). WIHS is a large, racially and geographically diverse cohort of HIV positive (n = 2761), and risk-matched HIV-negative women (n = 942). The large size of the cohort will provide substantial statistical power, which is of major importance in any HLA association study.

ELIGIBILITY:
* INCLUSION CRITERIA:

DNA and relevant clinical data from properly consented WIHS subjects (maximum estimated at 3500) will be provided to our lab for genotyping and analysis.

EXCLUSION CRITERIA:

No available subjects will be excluded.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3500 (Estimated)
Dates: Start 2002-07-15; Study Completion 2010-08-18

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Parham P, Ohta T. Population biology of antigen presentation by MHC class I molecules. Science. 1996 Apr 5;272(5258):67-74. doi: 10.1126/science.272.5258.67. PMID 8600539
- [Background] Hughes AL, Yeager M. Natural selection at major histocompatibility complex loci of vertebrates. Annu Rev Genet. 1998;32:415-35. doi: 10.1146/annurev.genet.32.1.415. PMID 9928486
- [Background] Carrington M, Nelson GW, Martin MP, Kissner T, Vlahov D, Goedert JJ, Kaslow R, Buchbinder S, Hoots K, O'Brien SJ. HLA and HIV-1: heterozygote advantage and B*35-Cw*04 disadvantage. Science. 1999 Mar 12;283(5408):1748-52. doi: 10.1126/science.283.5408.1748. PMID 10073943